CLINICAL TRIAL: NCT03913117
Title: Phase I Clinical Trial Assessing the Safety and Feasibility of Intramuscular pNGVL4aCRTE6E7L2 and TA-CIN Administration for the Treatment of Patients With Persistent HPV16+ ASC-US or LSIL
Brief Title: Study of Treatment for HPV16+ ASC-US or LSIL
Acronym: PVX-6
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rebecca Arend, Professor of Medicine, Division Director Gynecology Oncology, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB IND 18340; 000540585 (Other: John's Hopkins University)
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: ASC-US; LSIL
Keywords: HPV16
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- pNGVL4aCRTE6E7L2 0.3mg dose (Experimental): Low dose of pNGVL4aCRTE6E7L2 plasmid DNA is administered by intramuscular injection at weeks 0, 4 and 8.
  Interventions: Biological: pNGVL4aCRTE6E7L2
- pNGVL4aCRTE6E7L2 1 mg dose (Experimental): Intermediate dose of pNGVL4aCRTE6E7L2 plasmid DNA is administered by intramuscular injection at weeks 0, 4 and 8.
  Interventions: Biological: pNGVL4aCRTE6E7L2
- pNGVL4aCRTE6E7L2 3 mg dose (Experimental): High dose of pNGVL4aCRTE6E7L2 plasmid DNA is administered by intramuscular injection at weeks 0, 4 and 8.
  Interventions: Biological: pNGVL4aCRTE6E7L2
- PVX-6 (Experimental): Selected dose of pNGVL4aCRTE6E7L2 plasmid DNA is administered by intramuscular injection at weeks 0 and 4, and the TA-CIN protein is administered by intramuscular injection at week 8.
  Interventions: Biological: pNGVL4aCRTE6E7L2; Biological: TA-CIN

INTERVENTIONS:
Biological: pNGVL4aCRTE6E7L2 — Naked pNGVL4aCRTE6E7L2 DNA plasmid
Biological: TA-CIN — TA-CIN is a single fusion protein comprised of HPV16 L2, E7 and E6 proteins linked in tandem.
  Arms: PVX-6

SUMMARY:
Phase I clinical trial to assess safety of pNGVL4aCRTE6E7L2 DNA and TA-CIN protein vaccinations, and to seek the appropriate dose of the pNGVL4aCRTE6E7L2 DNA vaccine

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the safety and feasibility of intra-muscular administration of pNGVL4aCRTE6E7L2 DNA vaccine in patients with persistent HPV16+ ASC-US/LSIL.
2. To determine the appropriate intra-muscular injection dose of pNGVL4aCRTE6E7L2 DNA vaccine as determined by toxicity and immunogenicity for a subsequent phase II clinical trial.
3. To determine the safety and feasibility of intra-muscular administration of pNGVL4aCRTE6E7L2 DNA vaccine prime, TA-CIN protein vaccine boost in patients with persistent HPV16+ ASC-US/LSIL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent (>6 month period) ASC-US/LSIL determined by cervical cytology at study entry (ThinPrep with imaging)
2. Patients whose cytologic samples are persistent (>6 month period) HPV16+ by Roche Cobas 4800, Roche Linear Array HPV Genotyping test or other FDA-approved HPV genotyping test at study entry. Co-infections with HPV types other than HPV16 are permissible for study entry.
3. Age ≥ 19 years
4. Baseline Eastern Cooperative Oncology Group
5. Patients must have adequate organ function at the time of enrollment as defined by the following parameters:

   * White blood cell count > 3,000
   * Absolute lymphocyte number > 500
   * Absolute neutrophil count > 1,000
   * Platelets > 90,000
   * Hemoglobulin > 9
   * Total bilirubin <3 X the institutional limit of normal
   * AST(SGOT)/ALT(SGPT) <3 X the institutional limit of normal
   * Creatinine < 2.5X the institutional limit of normal
6. Women of child-bearing potential must agree to use two forms of contraception (hormonal and barrier) prior to study entry and for 3 months after study completion.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Subject is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patients with ASC-US/LSIL determined by cervical cytology at study entry that are HPV16 negative.
2. Histologic evidence of CIN2+
3. Patients with a diagnosis of immunosuppression or prolonged, active use of immunosuppressive medications such as steroids.
4. Prior vaccination with any HPV antigen (prophylactic or therapeutic).
5. Patients who are receiving any other investigational agents within 28 days prior to the first dose.
6. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with a history of autoimmune disease such as multiple sclerosis, exclusive of a history of thyroiditis, psoriasis, Sjrogen's, or inflammatory bowel disease.
8. Patients with a history of allergic reactions attributed to compounds used in agent preparation.
9. Patients who are pregnant or breast feeding.
10. Patient with active or chronic infection of HIV, HCV, or HBV.
11. Patients who have had a prior LEEP or cervical conization procedure.
12. History of prior malignancy permitted if patient has been disease free for ≥ 5 years; however individuals with completely resected basal cell or squamous cell carcinoma of the skin within this interval may be enrolled.
13. Inability to understand or unwillingness to sign an informed consent document.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with a cervical cytologic diagnosis of ASC-US or LSIL
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of pNGVL4aCRTE6E7L2 DNA vaccination | 12 months
  To determine the safety and feasibility of intra-muscular administration of pNGVL4aCRTE6E7L2 DNA vaccine in patients with persistent HPV16+ ASC-US/LSIL
Dose finding | 12 months
  To determine the appropriate intra-muscular injection dose of pNGVL4aCRTE6E7L2 DNA vaccine as determined by toxicity and immunogenicity for a subsequent phase II clinical trial
Safety and feasibility of PVX-6 vaccination | 12 months
  To determine the safety and feasibility of intra-muscular administration of pNGVL4aCRTE6E7L2 DNA vaccine prime, TA-CIN protein vaccine boost in patients with persistent HPV16+ ASC-US/LSIL

SECONDARY OUTCOMES:
HPV16 antibody response | 12 months
  To evaluate the levels of circulating antibody specific for HPV-16 in the peripheral blood pre- and post-vaccination
HPV16 CD8 T cell response | 12 months
  To evaluate the levels of circulating HPV-16 E6- and E7-specific CD8+ T cells and T regulatory cells in the peripheral blood pre- and post-vaccination
HPV16 L2E7E6 T cell proliferative response | 12 months
  To evaluate the proliferative responses of peripheral blood mononucleocytes pre- and post-vaccination in response to stimulation by HPV16 E6, E7 and L2
Clearance of HPV16 | 12 months
  To evaluate the presence of high risk HPV, and specifically HPV16 in cytologic specimens pre- and post-vaccination
Cytologic clearance | 12 months
  To evaluate changes in the cytopathology of ectocervical and endocervical specimens taken pre- and post-vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UAB | The University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland